CLINICAL TRIAL: NCT04303104
Title: A Randomized Controlled Trial to Evaluate a Scalable Active Case Finding Intervention for TB Using a Point-of-care Molecular Tool (Gene Xpert)
Brief Title: Xpert Active Case-finding Trial 3 (XACT-3)
Acronym: XACT-3
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: Zambart (University of Zambia), Zambia (Unknown); Instituto Nacional de Saúde, Mozambique (Other Government); Biomedical Research and Training Institute, Zimbabwe (Other); Radboud University Medical Center (Other); London School of Hygiene and Tropical Medicine (Other); University of Cape Town Lung Institute (Other)
Responsible Party: Principal Investigator, Keertan Dheda, Principal Investigator, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: XACT-3
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Tuberculosis
Keywords: TB Screening; Active Case Finding; Mobile versus Centralized
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Intervention Model Description: Xpert-oriented active case-fining model for TB: portable GXPU/molecular device hosted in a mobile mini-clinic to perform ACF in peri-urban informal settlements. Open-label randomisation to GXPU performed at POC or a central laboratory.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile ACF (Active Comparator): Xpert Edge performed at point-of-care employing a low-cost panel van that is staffed by three health care workers. Patients identified with active TB will be initiated on TB treatment on the same day at the nearest clinic. On site HIV testing will also be offered. Thus, the interventional package is one of ACF + POC TB testing (TB testing by Xpert will occur on site at the van).
  Interventions: Other: GeneXpert Edge
- Centralised ACF (Placebo Comparator): Similar to active arm but Xpert Ultra will be performed at a centralized laboratory (samples will be transported to the laboratory with results being available in a few days). Thus, the standard of care package is ACF + distant TB testing (TB testing by Xpert will occur at a distant laboratory site).
  Interventions: Other: GeneXpert Ultra

INTERVENTIONS:
Other: GeneXpert Edge — Screening intervention: novel diagnostic for Active Case Finding (GeneXpert MTB/RIF) for TB on sputum collected and performed at point-of-contact in a mobile van
  Arms: Mobile ACF
Other: GeneXpert Ultra — Screening intervention: novel diagnostic test for Active Case Finding (GeneXpert MTB/RIF) for TB on sputum collected at point-of-contact in a mobile van but sent to laboratory
  Arms: Centralised ACF

SUMMARY:
TB remains the foremost infectious disease killer globally. A startling statistic is that two out of every five TB cases globally (40%) remain undiagnosed and untreated. These 'missed' or undiagnosed cases are disproportionately concentrated in large peri-urban 'slums' and informal settlements of large cities in Africa and Asia (they are frequently minimally symptomatic but remain infectious).

The lack of a sensitive low cost same-day test represented a major challenge to active community-based case finding (ACF) compared to the current model where patients 'self-seek' care (passive case finding). More recently, sensitive TB DNA-detection tests called Gene Xpert (Xpert) have become available. This is a nucleic acid amplification test-based technology which can rule-in a diagnosis of TB in two thirds of smear negative pulmonary TB cases. GeneXpert® has now been rolled out in many African countries and is the frontline TB test in primary care clinics in South Africa. The investigators recently showed that GeneXpert® significantly reduced the time to treatment initiation in the setting of passive case finding (elaborated in next section). The investigators further showed that GeneXpert® can be performed by a minimally trained healthcare worker. However, historically technical and logistical demands meant that the GeneXpert® MTB-RIF assay was not ideally suited to use at point of care and in South Africa it is still centrally located.

Small portable battery-operated versions of these tests are now available (EDGE, GeneXpert two-module mobile platform). The investigators conducted a large study in South Africa and Zimbabwe (published in 2016) that showed that using the old non-portable version of Xpert on a mini-truck equipped with a generator was feasible and highly effective for ACF. A subsequent study funded by the American government (XACT II), showed that using the portable version of Xpert on the back of a small low-cost scalable panel van (in effect a mobile mini-clinic) was feasible and had a very high pick-up rate of TB in peri-urban communities (~10% of those undergoing targeted screening). In this study, the investigators will test the hypothesis that community-based active case finding (ACF) using Gene Xpert Edge (in a low cost scalable mini-mobile clinic) performed at point-of-care (POC) is feasible and more effective (lower proportion of TB cases failing to initiate treatment especially if they are 'super-spreaders' i.e. highly infectious) than Xpert performed in a centralised laboratory.

DETAILED DESCRIPTION:
In the proposed study (XACT III) the investigators will use the same approach (as for XACT II), but it remains to be shown that such a strategy is scalable and feasible in different settings where the challenges and conditions vary. More importantly, the investigators need to methodologically optimize the ACF model. Thus, the investigators aim to determine where Xpert (the diagnostic test) should be optimally placed from a physical location point-of-view, i.e. does it really need to be installed in the mobile mini clinic, or, can it be located in centralized laboratories (as it is now) with samples being sent to these laboratories? This is a very important question: it is known that sending collected sputum samples to centralized laboratories will be much easier as it uses existing infrastructure, however, the downside is between 20 and 40% of patients fail to come back to collect their results (pre-treatment loss to follow-up; PTLF). Using the diagnostic in the mobile mini van (at point-of-care; POC) dramatically reduces this PTLF enabling quick diagnosis and interrupting transmission. To definitively settle the question, a study is needed using the two different strategies to find out which strategy is most cost-effective yet can rapidly pick up the most cases and minimize transmission.

There are two other important sub-questions that the study will answer. Chest X-rays, which can identify people at high risk of having TB, can now be automatically read by a computer algorithm (called computer-assisted diagnosis of TB; CAD-TB). It will be very important to know whether mass screening using CAD-TB can triage individuals i.e. narrow the net so that the investigators target the ACF only to those at high risk of having TB. This could save even more money yet be just as effective.

Secondly, a fundamental unanswered question is why individuals with minimal or no symptoms can be highly infectious (transmit disease)? The investigators need to study this phenomenon in greater detail using cough aerosol readouts, chest X-rays, and looking at the TB strains. In addition the investigators would like to screen contacts of individuals with confirmed tuberculosis This might provide medical science with the information it needs to design diagnostic or therapeutic interventions to address this important problem.

However, the key priority now is to show that the XACT approach is feasible in different settings and to clarify how the molecular diagnostics should be optimally located. Answering these questions will allow the initiation of ACF programmes in many countries and will contribute critical data to policy makers so that guidelines on ACF can be disseminated and implemented.

ELIGIBILITY:
Inclusion Criteria:

1. Community participant willing to complete community-based symptom screening, finger-prick blood testing, and/or undergo TB diagnostic testing.
2. Provision of informed consent.
3. Has documentation of, or willingness to be tested for HIV infection. HIV testing does not need to be repeated if there is written documentation of a confirmed positive test at any time in the past.
4. HIV-negative adults (older than 18 years) with 1 or more of the following:• cough ≥ 2 weeks• loss of weight• Fever• night sweats• generalized fatigue• haemoptysis• chest pain.
5. Any HIV+ve adult (older than 18 years).
6. Agrees to the collection and storage of blood, urine, sputum specimens for use for future research. (The participant may decline collection of specimens for human genetic research and still be eligible for the study).

Exclusion Criteria:

1. Inability to provide informed consent (e.g. mentally impaired).
2. Patients who have completed TB treatment in the last 2 months, or who have self-presented to their local TB clinic and are currently being worked up for suspected TB.
3. Patients already diagnosed with active TB.
4. Patients unable to commit to a two month follow up or who do not wish to be followed up.

Inclusion criteria for Household contacts (HHC)

1. Adult (> 18 years old) with significant recent exposure (within the past 6 months) to an adult with untreated or inadequately treated pulmonary TB.
2. No clinical signs or symptoms of active TB that include, but are not limited to: persistent cough, haemoptysis, fever, unintended weight loss or failure to thrive (children), fatigue or lethargy, night sweats, pleuritic chest pain, draining lymph node, or other evidence of extra-pulmonaryTB. If clinical signs or symptoms of TB are present, Chest X-Ray and/or sputum culture results must be included in the overall evaluation to rule out active TB.
3. Has signed a written consent or witnessed oral consent in the case of illiteracy, prior to his/her first sample or other study-specific data being collected.
4. Agrees to the collection and storage of blood, urine, saliva and sputum specimens for use for future research. (The participant may decline collection of specimens for human genetic research and still be eligible for the study.)

Exclusion Criteria for Household contacts

1. Plans to move from his/her current residence, which would interfere with the participant's ability to complete all study visits (through the Month 24Visit).
2. Has an active psychiatric condition, or alcohol or drug dependence that, in the opinion of the site investigator or designee, might interfere with the ability to give true informed consent and to adhere to the study requirements.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3394 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion with PTLF (defined as test positive patients failing to initiate treatment by 60 days) and/ or the proportion of infectious TB patients (smear positive and/ or with cavitatory disease) not initiating treatment within 14 days of diagnosis. | Within 2 months of enrollment, up to 24 months
  The proposed primary outcome measure is a surrogate of transmission and disease amplification (especially of the 'missed' highly infectious cases). Thus, the composite outcome serves as a surrogate of those who will experience a poor outcome (the missing cases) and disease amplification (transmission of TB).

SECONDARY OUTCOMES:
Proportion of culture-positive patients failing to initiate treatment in each study arm within 14 days of diagnosis. | Within 2 months of enrolment, up to 26 months
  Proportion of culture-positive participants not initiating treatment as confirmed by TB Clinic attendance register.
Time to TB treatment initiation | Within 2 months of enrollment, up to 24 months
  Time (in days) as determined by difference between enrollment date and date that treatment is commenced in local TB Clinic as per attendance register.
Time-specific proportion of patients initiated on TB treatment up to 60 days. | Within 2 months of enrolment, up to 26 months
  Proportion of culture-positive participants initiating treatment as confirmed by TB Clinic attendance register.
Feasibility of Xpert being performed by minimally trained health care workers at point-of-care using. | Through study completion, up to 48 months
  Number of study days lost to operational problems with machine or van (recorded daily by study team in daily register). Furthermore, user adherence to test protocol, operator knowledge of the testing procedure, and confidence in the test and satisfaction with its ease of use will be tested by two standardized questionnaires employed and validated in our previous study on active case-finding using lab-based Xpert.
Cost effectiveness analysis in each of the four countries. | Through study completion, up to 48 months
  Cost-effectiveness analysis to be performed at study conclusion.
Turn-around-time for Xpert testing in both arms. | Within 2 months of enrolment, up to 26 months
  Number of days wait until dispatch of result to patient.
Transmission impact using modelling based on exposure scores, imaging and CASS. | Within 2 months of enrolment, up to 26 months
  This is a composite outcome determined by individual score for each of the mechanisms (contact, imaging and CASS) used to investigate transmission.
Household contact tracing yield from TB positive patients (active TB and QFT conversion). | Within 2 months of enrolment, up to 26 months
  Captured as number of TB positive contacts for an enrolled participant with active TB.
The time-specific proportion of culture-positive TB cases initiating TB treatment in each study arm. | Through study completion, up to 48 months
  Number of culture confirmed cases who initiate treatment in each arm.
The proportion of culture-positive TB cases completing 6-months of TB treatment in each study arm. | Within 8 months of enrolment, up to 48 months
  Number of culture confirmed cases who initiate treatment in each arm and finish the course as per TB clinic register.

CONTACTS AND LOCATIONS:
Overall Officials: Keertan Dheda, MBChB, PhD, Principal Investigator — Lung Infection and Immunity Unit and Division of Pulmonology
Locations (4):
- Bindiya Meggi, Maputo, Mozambique
- University of Cape Town, Cape Town, Western Cape, South Africa
- Helen Ayles, Lusaka, Zambia
- Junior Mutsvangwa, Harare, Zimbabwe